CLINICAL TRIAL: NCT02570802
Title: Ultrasonographic Reference Values for Peripheral Nerves and Nerve Roots in the Normal Population of Children and Adolescents
Brief Title: Ultrasonographic Reference Values for Peripheral Nerves in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Nerve US Children 01
Record Dates: First submitted 2015-09-14; First posted 2015-10-07 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Normal Values of Peripheral Nerves in Healthy Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasound of peripheral nerves (Other): Ultrasonographic examination
  Interventions: Procedure: Ultrasonographic examination

INTERVENTIONS:
Procedure: Ultrasonographic examination

SUMMARY:
The purpose of this clinical trial is to assess normal values of the cross-sectional area of peripheral nerves and nerve roots in children and adolescents between 2 and 18 years.

DETAILED DESCRIPTION:
This is a single center prospective clinical trial to determine standard values of the cross-sectional area of the median, ulnar, radial, peroneal, tibial, sural and vagus nerve as well as C5, C6 and C7 cervical roots in a cohort of neuromuscular unaffected children and adolescents between 2 and 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between 2 and 18 years
* Written informed consent of the caregivers and the children/adolescents between 14 and 18 years

Exclusion Criteria:

* Inability to meet study requirements
* Neuromuscular disease or symptoms

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 255 (Estimated)
Dates: Start 2015-10; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional area (mm2) of the C5 cervical root in children and adolescents from 2 to 18 years | one year
  Cross-sectional area will be displayed as percentiles according age, weight and length
Cross-sectional area (mm2) of the C6 cervical root in children and adolescents from 2 to 18 years | one year
  Cross-sectional area will be displayed as percentiles according age, weight and length
Cross-sectional area (mm2) of the C7 cervical root in children and adolescents from 2 to 18 years | one year
  Cross-sectional area will be displayed as percentiles according age, weight and length
Cross-sectional area (mm2) of the radial nerve in children and adolescents from 2 to 18 years | one year
  Cross-sectional area will be displayed as percentiles according age, weight and length
Cross-sectional area (mm2) of the superficial radial nerve in children and adolescents from 2 to 18 years | one year
  Cross-sectional area will be displayed as percentiles according age, weight and length
Cross-sectional area (mm2) of the peroneal nerve in children and adolescents from 2 to 18 years | one year
  Cross-sectional area will be displayed as percentiles according age, weight and length
Cross-sectional area (mm2) of the tibial nerve in children and adolescents from 2 to 18 years | one year
  Cross-sectional area will be displayed as percentiles according age, weight and length
Cross-sectional area (mm2) of the sural nerve in children and adolescents from 2 to 18 years | one year
  Cross-sectional area will be displayed as percentiles according age, weight and length
Cross-sectional area (mm2) of the vagus nerve in children and adolescents from 2 to 18 years | one year
  Cross-sectional area will be displayed as percentiles according age, weight and length

SECONDARY OUTCOMES:
Interrater reliability | one year
  Reliability is expressed by the intraclass correlation coefficient (ICC)
Intrarater reliability | one year
  Reliability is expressed by the intraclass correlation coefficient (ICC)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Fischer, MD, Principal Investigator — University of Basel, Children's Hospital
Locations (1):
- University of Basel, Children's Hospital, Basel, Switzerland

REFERENCES:
- [Derived] Rasenack M, Decard BF, Schadelin S, Grimm A, Fischer D, Hafner P. Ultrasonographic reference values for peripheral nerves and nerve roots in the normal population of children and adolescents: study protocol for an observational-prospective trial. BMJ Open. 2016 Dec 9;6(12):e014662. doi: 10.1136/bmjopen-2016-014662. PMID 27940636